CLINICAL TRIAL: NCT04946357
Title: Neoadjuvant Irradiation of Extremity Soft Tissue Sarcoma With Ions
Acronym: EXTREM ION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXTREM ION
Record Dates: First submitted 2021-06-21; First posted 2021-06-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Protons, 39 Gy (RBE) in 13 fractions (single dose 3.0 Gy(RBE)) (Experimental): Arm A: Protons, 39 Gy (RBE) in 13 fractions (single dose 3.0 Gy(RBE))
  Interventions: Radiation: Protons
- Arm B: Carbon ions, 39 Gy(RBE) in 13 fractions (single dose 3.0 Gy(RBE)) (Experimental): Arm B: Carbon ions, 39 Gy(RBE) in 13 fractions (single dose 3.0 Gy(RBE))
  Interventions: Radiation: carbon ions

INTERVENTIONS:
Radiation: Protons — proton irradiation with a total dose of 39 Gy(RBE) in 3 Gy(RBE) fractions
  Arms: Arm A: Protons, 39 Gy (RBE) in 13 fractions (single dose 3.0 Gy(RBE))
Radiation: carbon ions — carbon ion irradiation with a total dose of 39 Gy(RBE) in 3 Gy(RBE) fractions
  Arms: Arm B: Carbon ions, 39 Gy(RBE) in 13 fractions (single dose 3.0 Gy(RBE))

SUMMARY:
This randomized prospective open-label phase 2 trial testes the safety and feasibility of a hypofractionated accelerated neoadjuvant proton or carbon ion radiotherapy based on the rate of wound healing disorders from beginning of radiotherapy to maximum 120 days after the planned tumor resection or discontinuation of treatment due to any reason. The treatment is of shorter duration (2-3 weeks vs. 5 weeks standard treatment), which should please most patients and thus enhance quality of life. The treatment regimen furthermore promises a reduced rate of late side effects and significant optimization of the current treatment standards. A phase II trial is mandatory not only for obtaining the safety and feasibility data, but also in order to prepare a concurrent phase III trial. Due to the low incidence of soft tissue sarcoma, only a well prepared multicenter study has a chance to be successfully completed based on previous experiences in trials for seldom tumor entities.

DETAILED DESCRIPTION:
Oncologic complete local excision (wide resection) combined with radiotherapy forms the standard treatment for patients with soft tissue sarcoma. Especially patients with G2/G3 sarcomas profit from the combination of radiotherapy and surgery. Well-differentiated sarcomas (G1) after total resection (R0) receive no subsequent treatment besides surgery. The sequence of surgery and radiation therapy is widely discussed by the radiation oncologists and surgeons. The main advantages of neoadjuvant (pre-operative) radiotherapy are the smaller treatment target volumes and reduced prescribed radiation doses of 50 Gy vs. 66 Gy (postoperative) in 2 Gy single doses. Thus, due to these reductions in volumes and dose, neoadjuvant radiotherapy is associated with a lower rate of radiotherapy-associated edema and fibrosis. However, a randomized phase III study showed an increased rate of wound healing complications in patients with neoadjuvant radiotherapy compared to adjuvant (post-operative) radiotherapy (35% vs. 17%). For this reason, adjuvant radiotherapy in is currently preferred in cases with good operability.

Particle therapy bears the chance to utilize the advantages of preoperative radiotherapy without compromising wound healing. The advantages of tumor treatment by ion therapy are based on their special biological and physical features. Protons and carbons ion lead to an improved dose distribution compared to photons which allows an improved sparing of the neighboring risk organs and at the same time an escalation of the dose prescribed to the tumor. Carbon ions are furthermore superior to protons by biological advantages based on their enhanced biological effectivity. In general, heavy ions are considered as a good treatment option for tumors of low radiosensitivity as sarcomas. Superior survival and decreased toxicity rates are expected from the use of protons and carbon ions.

This randomized prospective open-label phase 2 trial testes the safety and feasibility of a hypofractionated accelerated neoadjuvant proton or carbon ion radiotherapy based on the rate of wound healing disorders from beginning of radiotherapy to maximum 120 days after the planned tumor resection or discontinuation of treatment due to any reason. The treatment is of shorter duration (2-3 weeks vs. 5 weeks standard treatment), which should please most patients and thus enhance quality of life. The treatment regimen furthermore promises a reduced rate of late side effects and significant optimization of the current treatment standards. A phase II trial is mandatory not only for obtaining the safety and feasibility data, but also in order to prepare a concurrent phase III trial. Due to the low incidence of soft tissue sarcoma, only a well prepared multicenter study has a chance to be successfully completed based on previous experiences in trials for seldom tumor entities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed soft-tissue sarcoma of the extremities with an indication for perioperative radiation treatment
* Resectable or marginally resectable
* Karnofsky index of ≥ 70%
* Age ≥ 18 years
* Carried out patient education and written consent
* Patient is capable to give informed consent

Exclusion Criteria:

* Stage IV (distant metastases)
* Lymph node metastasis
* Metal implants that influence treatment planning with ions
* Previous radiotherapy in the treatment area
* Desmoid tumors
* Simultaneous participation in another clinical trial that could influence the results of the study.
* Active medical implants for which no ion beam irradiation permit exists at the time of treatment (e.g., cardiac pacemaker, defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of therapies without wound healing disorders and/or discontinuation | from the beginning of radiotherapy (day1) until a maximum of 120 days after the resection
  Proportion of therapies without wound healing disorders and / or discontinuation in each study arm.

SECONDARY OUTCOMES:
LC: Local control | from start of radiotherapy to local onset to local tumor progression up to 5 years
  LC: Local control determined from local onset to local tumor progression
LPFS: locally progression-free survival determined from onset of therapy to local tumor progression | from start of radiotherapy to onset of therapy of local tumor progression up to 5 years
  LPFS: locally progression-free survival determined from onset of therapy to local tumor progression
DFS: Disease-free survival | from start of radiotherapy to onset of therapy until local and / or distant tumor progression up to 5 years
  DFS: Disease-free survival determined from onset of therapy until local and / or distant tumor progression
OS: Overall survival | from start of radiotherapy until death or censorship up to 5 years
  OS: Overall survival until death or censorship

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Department of RadioOncology, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brugemann D, Lehner B, Kieser M, Krisam J, Hommertgen A, Jaekel C, Harrabi SB, Herfarth K, Mechtesheimer G, Sedlaczek O, Egerer G, Geisbusch A, Uhl M, Debus J, Seidensaal K. Neoadjuvant irradiation of extremity soft tissue sarcoma with ions (Extrem-ion): study protocol for a randomized phase II pilot trial. BMC Cancer. 2022 May 12;22(1):538. doi: 10.1186/s12885-022-09560-x. PMID 35550036